CLINICAL TRIAL: NCT04576442
Title: Evaluation of the Asthma Management Program to Promote Activity for Students in Schools (Asthma-PASS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: University of Rochester (Other); Columbia University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-10930; R33HL147908 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma-PASS Intervention (Experimental): Collaboration with PCPs to optimize management. Community Health Worker (CHW) to ensure PCP plan is followed. Two asthma education sessions with children/caregivers focusing on self-efficacy and physical activity promotion. Promotion of asthma awareness in school. School personnel training in asthma
  Interventions: Behavioral: Asthma-PASS; Behavioral: Child/Caregiver Education session
- Asthma Management Comparison Group (Active Comparator): Includes two sessions of basic asthma education and PCP notification of child's asthma severity level.
  Interventions: Behavioral: Basic Asthma Management (AM); Behavioral: Child/Caregiver Education session

INTERVENTIONS:
Behavioral: Asthma-PASS — The investigator will collaborate with the student's primary care provider (PCP) by sending a letter via facsimile, and/or email to ensure appropriate medications are prescribed or adjusted and rescue medications are available at school. Community Health Workers (CHWs) will follow up with PCPs as needed to provide reminders about prescriptions for controlled medications and to ensure a MAF is provided to schools to allow rescue medication administration by nurses. CHWs will work with local pharmacies when possible to have prescribed medications delivered to schools and homes. For students without a PCP, we will refer families to one of Montefiore Medical Center's 20 practices throughout the Bronx. For students without medical insurance or who are unable to go to a Montefiore clinic, the NYC DOE physicians who routinely attend NYC schools will provide medical care and prescribe appropriate medications.
  Arms: Asthma-PASS Intervention
Behavioral: Basic Asthma Management (AM) — PCPs and caregivers will be notified that children in the AM group have persistent/uncontrolled asthma that warrants use of guideline-based preventative medications.
  Arms: Asthma Management Comparison Group
Behavioral: Child/Caregiver Education session — The investigator will provide in-school child asthma education sessions delivered by trained, bilingual (English-Spanish) Community Health Workers (CHWs) using an established manualized protocol from past and current studies designed to improve knowledge and self-efficacy. Each child will receive two 1-on 1, 20-minute developmentally appropriate educational sessions at school 3-4 weeks apart. Sessions will cover: 1) asthma basics, symptoms and triggers; and 2) medications and correct administration technique. Caregivers will be called after each child session to highlight key points reviewed with the child and answer questions.

SUMMARY:
Physical activity (PA) is an important component of asthma management in children. Studies show that PA is associated with decreased severity of asthma symptoms, as well as improved disease control and quality of life. However, urban minority children with asthma face barriers to PA on multiple levels.The goal of this research project is to evaluate whether a multifaceted school-based intervention that addresses key barriers to physical activity reduces asthma morbidity among urban schoolchildren with asthma.

DETAILED DESCRIPTION:
Investigators will conduct a cluster-randomized controlled trial with 416 children ages 5-11 years with persistent or uncontrolled asthma from 26 Bronx schools. Schools will be randomly assigned to either (1) the Asthma-PASS intervention or an asthma management (AM) comparison group. Both groups will participate in an existing classroom-based daily activity program. Enrollment will occur over 4 consecutive school years with 6-8 schools joining the study each year. The investigators will assess the effectiveness of Asthma-PASS in reducing asthma morbidity, and improving PA as well as additional clinical and functional outcomes. The investigators will also identify potential mediators and moderators of the intervention effect. They will evaluate the process of intervention implementation by applying the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma (based on parent report with validation from the child's physician).
* Mild persistent or more severe asthma, or asthma that is uncontrolled despite therapy
* Attending kindergarten through 5th grade in Bronx elementary schools
* Parent is able to speak and understand either English or Spanish.
* Consent from the primary caregiver, caregiver permission for child participation as well as assent from the child (for age 7 and above).

Exclusion Criteria:

* No access to a phone to conduct follow-up surveys.
* Family plans to leave the school or city in less than 6 months.
* The child has other significant medical conditions, such as congenital heart disease, cystic fibrosis, or other chronic lung disease.
* Child is unable to participate in routine PE classes as per physician-completed sports participation form.
* Children in foster care or other situations in which consent cannot be obtained from a guardian.
* Child is a participant in a concurrent asthma intervention study.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in the number of Symptom free days (SFDs) | Baseline, 3, 6, 9, and 12 months
  Change from baseline in the number of SFDs will be assessed. Caregivers will report the number of days their child experienced no symptoms of asthma (defined as 24 hours with no coughing, wheezing, chest tightness, or shortness of breath) over the prior 14 day period. Symptom diaries provided as part of the study will be used to assist with recall. The trial will be successful if the intervention demonstrates a significantly greater improvement over time on SFDs at any of the 4 post-baseline assessments.

SECONDARY OUTCOMES:
Physical activity | Baseline, 3, 6 and 9 months
  Physical activity will be assessed by the number of minutes the child engages in 'moderate-vigorous' physical activity based on measurements taken using the ActiGraph GT3X+ activity monitor, a small, tri-axial micro-electromechanical system (MEMS) based accelerometer. Measurements will be taken over 7 consecutive days at baseline, 3, 6 and 9 months using the activity monitor. Children will wear the monitor on their waist, secured using an elastic belt. The number of minutes the child is in 'moderate-vigorous' physical activity will be summarized by study arm.

OTHER OUTCOMES:
Pediatric Asthma Caregiver's Quality of Life | 3-12 months
  Validated caregiver asthma related quality of life survey; 13 items, 7-point scale (ranging from 1-7); higher score indicates less impairment
Childhood Asthma Control Test | 3-12 months
  asthma control based on symptom frequency; score 0-27; higher score indicates well controlled asthma; score 19 or less indicates uncontrolled asthma.
Adherence | 3-12 months
  controller medication adherence, score range 0-4; higher scores corresponding to recommended behavior.
Asthma self-management questionnaire | 3-12 months
  caregiver self-management behavior; score range 0-100; higher score indicates more knowledge of self-management
Asthma knowledge | 3-12 months
  Caregiver asthma knowledge using sub-scale of Asthma Illness Representation Scale; score range 1-5; higher score represent better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No